CLINICAL TRIAL: NCT06495827
Title: Zhongshan Hospital，Fudan University
Brief Title: Predicting Response to Chemotherapy in Colorectal Cancer Via Multi-dimensional Analyses of the Tumor Associated Neutrophils
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of colorectal surgery department, Principal Investigator, Clinical Professor, Zhongshan Hospital, Fudan University
Other Study IDs: TANs for CT response in CRC
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Tumor Associated Neutrophils

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- response cohort: CRC patients with response status after chemotherapy
  Interventions: Other: No different intenvention
- resistance cohort: CRC patients with resistance status after chemotherapy
  Interventions: Other: No different intenvention

INTERVENTIONS:
Other: No different intenvention — No different intenvention

SUMMARY:
A single biomarker is not adequate to identify patients with colorectal cancer (CRC) who have the potential to benefit from adjuvant therapy, presumably owing to the complexity of tumor-infiltrating immune cells (TIICs). The density and spatial organization of TIICs has not been definitely established to explore their predictive value. This study aimed to investigate the prognostic significance of TIICs and its biological predictive value in CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written ICF.
2. The Eastern Cancer Collaborative Organization (ECOG) has a physical fitness score of 0 or 1.
3. The expected survival period is ≥ 3 months.

5. Subjects diagnosed with metastatic colorectal adenocarcinoma by histology or cytology.

6. Colorectal cancer patients who have not received systematic anti-tumor therapy in the past.

Exclusion Criteria:

1. Subjects suffered from other malignant tumors within 3 years before enrollment, except for cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, etc.).
2. Simultaneously enroll in another clinical study, unless it is an observational, non-interference clinical study or a follow-up period of an intervention study.
3. Received systematic anti-tumor therapy (chemotherapy) within 3 weeks prior to the first administration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled multiple cohorts, consisting of 653 tumor microarray specimens of CRC patients from Zhongshan Hospital
Sampling Method: Non-Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
PFS | From date of operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  From date of operation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months

IPD SHARING:
Plan to Share IPD: No